CLINICAL TRIAL: NCT02667652
Title: The Curative Effect of the Length of the Jejunum Exclusion in Grstric Bypass Surgery for Type 2 Diabetes:a Randomized Controlled Trials
Brief Title: The Curative Effect of the Length of the Jejunum Exclusion in Grstric Bypass Surgery for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weidong Tong (Other)
Responsible Party: Sponsor-Investigator, Weidong Tong, Gastric & Colorectal Division, General Surgery Dept. Daping Hospital, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 776117
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: T2DM; RYGB; RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- short biliarypancreatic limb (Active Comparator): short biliarypancreatic limb
  Interventions: Procedure: short biliarypancreatic limb
- long biliarypancreatic limb (Active Comparator): long biliarypancreatic limb
  Interventions: Procedure: long biliarypancreatic limb

INTERVENTIONS:
Procedure: short biliarypancreatic limb — biliarypancreatic limb:50cm;roux limb:150cm.
  Arms: short biliarypancreatic limb
Procedure: long biliarypancreatic limb — biliarypancreatic limb:100cm;roux limb:100cm.
  Arms: long biliarypancreatic limb

SUMMARY:
The purpose of this study is to investigate the curative effect of the length of the jejunum exclusion in gastric surgry for T2DM and metabolic syndrome,and to draft Scientific and reasonable operation parameters.

DETAILED DESCRIPTION:
Currently, there is a growing evidence supports the efficacy of Roux-en-Y gastric bypass for the treatment of Type 2 diabetes mellitus. However,there still have a great controversy about the operation parameters. With randomized controlled trial, Patients of BMI>21kg/m2 with type 2 diabetes were randomly divided into two groups: short biliarypancreatic limb:50cm;long biliarypancreatic limb :100cm. The investigators followed-up 3,6,12,24 months of the change of BMI,FBG,HbA1c,Blood pressure,Blood fat after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years old
* History of diabetes is less than 15 years
* Fasting c-peptide≥1.6
* BMI≥21kg/m2；
* Ability to understand the nature of the procedure and willing to follow postoperative routine lifestyle and checkups

Exclusion Criteria:

* Psychological and mental disorders
* Serious important organs such as heart and lung disease cannot be tolerated surgery
* Complex history of abdominal surgery in the abdominal cavity adhesion
* Pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
body mass idex | 24 months
  Changesd of BMI

SECONDARY OUTCOMES:
IFG | 24 months
  Variations of IFG
HbA1c | 24 months
  The changes of HbA1c
blood pressure | 24 months
  Changes of blood pressure including both systolic and diastolic pressure.
blood fat | 24 months
  Changes of blood fat including LDL, HDL, CHOL, TG

CONTACTS AND LOCATIONS:
Overall Officials: Tong Weidong, Professor, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Ethics Committee of Daping Hospital

REFERENCES:
- [Background] Shi Z. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Jun 24;362(25):2425; author reply 2426. doi: 10.1056/NEJMc1004671. No abstract available. PMID 20573933
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Gleysteen JJ. Five-year outcome with gastric bypass: Roux limb length makes a difference. Surg Obes Relat Dis. 2009 Mar-Apr;5(2):242-7; discussion 247-9. doi: 10.1016/j.soard.2008.08.005. Epub 2008 Aug 19. PMID 18996751
- [Background] Huang CK, Lee YC, Hung CM, Chen YS, Tai CM. Laparoscopic Roux-en-Y gastric bypass for morbidly obese Chinese patients: learning curve, advocacy and complications. Obes Surg. 2008 Jul;18(7):776-81. doi: 10.1007/s11695-007-9373-y. Epub 2008 May 16. PMID 18483835